CLINICAL TRIAL: NCT04287634
Title: Comparison Between the Segmental Mobilization and Entire Segmental Spine Mobilization in Cervical Spondylosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Kiran REC-00296
Record Dates: First submitted 2020-02-25; First posted 2020-02-27 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Cervical Spondylosis
MeSH Terms: conditions — Spondylosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Segmental Mobilization (Experimental): Hot Fermentation Soft tissue mobilization + Targeted Segmental Mobilization Home plan exercise= cervical muscles stretching, postural care
  Interventions: Other: Segmental Mobilization
- Entire Spine Mobilization (Experimental): Hot fermentation Soft tissue mobilization + Entire spine mobilization Home plan exercises=cervical muscles stretches, postural care
  Interventions: Other: Entire Spine Mobilization

INTERVENTIONS:
Other: Segmental Mobilization — Hot fermentation =10 minutes Soft tissue mobilization =5 minutes Targeted segmental mobilization= 3 sets of 10 repetitions Home plan exercise= cervical muscles stretching, postural care.
  Arms: Segmental Mobilization
Other: Entire Spine Mobilization — Hot fermentation=10 minutes Soft tissue mobilization=5 minutes Entire spine mobilization =3 sets of 10 repetitions Home plan exercises=cervical muscles stretches, postural care.
  Arms: Entire Spine Mobilization

SUMMARY:
All the patients of cervical spondylosis which were enrolled in this study were assessed in Rehabilitation centre of Yusra General Hospital. Patients who compete the inclusion criteria are randomly assigned by the seal envelop method in to two groups interventional and control group. There is nine sessions of three weeks rehabilitation program and Pain is assessed on Numeric pain rating scale, Disability on Neck Disability index and ROM is assessed by Goniometer in 1ST, 4TH and last visit. Three sessions of intervention is given to patient per week.

DETAILED DESCRIPTION:
Cervical spondylosis which is the common age related process having disturbing one or multiple segments of cervical spine. Cervical spondylosis shows a series of changes that is degenerative changes of discs and facet joints including bony growths of bodies of vertebrae, hypertrophy of arches of lamina and facet joints and instability of various segments in cervical spine. Origin of any degenerative disorders is linked with aging process. Cervical spondylosis worsens with age.As the age increases the cartilages and bones that make up our spine gradually develop wear and tear these changes can include dehydrated discs, herniated discs, bony spurs and causes neck injuries.

Mechanical neck disorders will great react to conservative management, but the gold standard intervention for the mechanical neck pain has yet to be recognized. There are many interventions which have Some treatments have been review in various randomized control studies (RCT), but I will show the best accessible evidence for the mostly common used ones.

Conservative management of the neck pain is respond well .On daily activities postural awareness and stress management strategies, work place (ergonomics) or hobbies may be valuable in many patients. Patient reeducation is necessary and advised to patient to use merely one pillow at night and When the intensity of pain is high, anti- inflammatory agents or analgesics are broadly and commonly used. Tricycle antidepressants having low dose for example amitriptyline( 10-30 mg) each night, may produce better results .Yoga ,Alexander techniques and pilates exercises are essential for improving posture of neck but the cost of these interventions in treating pain in neck is tentative.

Randomized controlled studies (RCT) which is included in meta analysis of Manual therapy interventions therapy (Manipulation or mobilization physiotherapy ) provide inadequate evidence that mobilization techniques and manipulation are more valuable for the treatment of the severe neck pain as compared to the active treatments (patient reeducation, counseling, drug therapy ). However, manipulation as compared to mobilization has been linked with severe neurological complications and damages round about 5-10 per 10 million manipulations.

Manipulation (high velocity amplitude thrust ), Mobilization or therapeutic exercises appear to be equally successful . A study which evaluate manipulation with therapeutic exercise whether modality separately used proved the combination to be more valuable for three months but there is no significant difference was notice than the exercises therapy only from one to two years . However, one more study showed no significant advantage for six weeks and six months by additional interventions manual therapy techniques, mobilization physiotherapy of 63% of population or shortwave diathermy(SWD) along with exercise and advice.

Meta analysis of various frail randomized controlled trials and studies showed no strong evidence about the value ability and usefulness of both manual and mechanical traction and acupuncture with a range of other treatments in patients with chronic pain in neck. Further additional interventions techniques like psychotherapy for example cognitive behavioral therapy also cause extra and additional effects to mechanical and physical intervention alone. Many studies and systemic reviews are required to evaluate the effectiveness and usefulness of standardized interventions in patients of cervical spondylosis. Due to finding the long term effects the lengthy follow up of interventions , large sample size ,lack of regularity in study designs and using multiple set up across the studies are complicated. Analyses will also be tough because of the use of more than one intervention strategies in same study design.Strong evidences are required to identify the cost effectiveness of intervention strategies.

A study on identify the effects of central and unilateral posterior anterior (UPA) mobilization technique on cervical spine lordosis, stiffness of muscles and range of motion in cervical spondylosis .There were significant Improvement in Cervical lordosis .however Muscle stiffness was significantly reduce after intervention and the effect of treatment lasted for five days without any supplementary intervention. The angles of cervical flexion and cervical extension angles were greater than before. Both the angles of lateral flexion and left rotation were significantly better and the effects of treatment which is proceeding for five days without any extra intervention. These results suggests that central and UPA mobilization manual therapy techniques is more valuable and effective in increasing cervical lordosis and range of motion, and lessening of stiffness of muscles in patients having cervical spondylosis.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of Cervical Spondylosis more than month
* Limited Cervical ROM (at least any 2 ROM)

Exclusion Criteria:

* Positive Vertebrobasilar Insufficiency & Sharp Purser Test
* Spinal stenosis.
* Osteoporosis.
* Trauma.
* Spondylosis
* Inflammatory arthritis.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-07-14 (Actual)

PRIMARY OUTCOMES:
Neck Disability Index | 3 Week
  Neck Disability Index is the patient completed, specific condition related functional questionnaire with scoring 10 item that is pain, lifting, personal care, headaches, driving, concentration , recreation, work, reading and sleeping. Neck Disability Index can be used for musculoskeletal neck pain having chronic (more than 3 months), whiplash linked disorders and cervical radiculopathy. The neck disability index is translated in various languages having its own reliability and validity. In every 10 items scores, Activities of daily living (ADLs) are linked to 7 scores, 2 scores are associated to pain and 1 score are correlated to concentration. The scores from every item ranges from 0 to 5 and the final score is reported in percentage with total likely score is 100%
Numeric Pain Rating Scale (NPRS) | 3 Week
  NPRS numeric scale ranges from 0 to 10 in which no pain is shows by 0 point and worst pain is showed by 10 point, the pain explain as worst as you can .
Range of Motion (ROM) of cervical spine | 3 Week
  Changes from the Baseline, Goniometer was used to measure Cervical Range of motion. For determine ROM of cervical spine, the patients were ask to sit straight with their thoracic area supported with a back of a chair. Patient's feet were placed horizontally on the floor with knees and hips at right angle to each other and arms were folded over the chest to reduce movement in the thoracic region. The patients were asked to move the head as far as possible in a standard manner. All the ranges of cervical spine that is flexion, extension, right and left side bending, and right and left side rotation is measured.

CONTACTS AND LOCATIONS:
Overall Officials: Abdul Ghafoor Sajjad, Phd*, Principal Investigator — Riphah International University
Locations (1):
- Yusra General Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Celenay ST, Akbayrak T, Kaya DO. A Comparison of the Effects of Stabilization Exercises Plus Manual Therapy to Those of Stabilization Exercises Alone in Patients With Nonspecific Mechanical Neck Pain: A Randomized Clinical Trial. J Orthop Sports Phys Ther. 2016 Feb;46(2):44-55. doi: 10.2519/jospt.2016.5979. Epub 2016 Jan 11. PMID 26755405
- [Background] Langevin P, Desmeules F, Lamothe M, Robitaille S, Roy JS. Comparison of 2 manual therapy and exercise protocols for cervical radiculopathy: a randomized clinical trial evaluating short-term effects. J Orthop Sports Phys Ther. 2015 Jan;45(1):4-17. doi: 10.2519/jospt.2015.5211. PMID 25420010
- [Background] Boyles R, Toy P, Mellon J Jr, Hayes M, Hammer B. Effectiveness of manual physical therapy in the treatment of cervical radiculopathy: a systematic review. J Man Manip Ther. 2011 Aug;19(3):135-42. doi: 10.1179/2042618611Y.0000000011. PMID 22851876
- [Background] Kanlayanaphotporn R, Chiradejnant A, Vachalathiti R. Immediate effects of the central posteroanterior mobilization technique on pain and range of motion in patients with mechanical neck pain. Disabil Rehabil. 2010;32(8):622-8. doi: 10.3109/09638280903204716. PMID 20205574
- [Background] Forbush SW, Cox T, Wilson E. Treatment of patients with degenerative cervical radiculopathy using a multimodal conservative approach in a geriatric population: a case series. J Orthop Sports Phys Ther. 2011 Oct;41(10):723-33. doi: 10.2519/jospt.2011.3592. Epub 2011 Sep 4. PMID 21891879